CLINICAL TRIAL: NCT06147635
Title: Prophylactic Tributyrin Supplementation in Acute Pancreatitis; a Phase IIa (Proof of Concept) Double-blind Randomized Placebo-controlled Food Supplement Trial
Brief Title: Prophylactic Tributyrin Supplementation in Acute Pancreatitis
Acronym: PARROT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, HC van Santvoort, dr. prof., St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL81496.100.22
Record Dates: First submitted 2023-07-10; First posted 2023-11-27 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-02

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Micro-encapsulated tributyrin granules, 4 grams three times daily, for a maximum of 14 days
  Interventions: Dietary Supplement: Micro-encapsulated granules of tributyrin (intervention)
- Control group (Placebo Comparator): Micro-encapsulated sunflower oil granules, 4 grams three times daily, for a maximum of 14 days
  Interventions: Dietary Supplement: Micro-encapsulated granules of sunflower oil (placebo)

INTERVENTIONS:
Dietary Supplement: Micro-encapsulated granules of tributyrin (intervention) — Three times daily 4 grams of micro-encapsulated granules of tributyrin, for a maximum of 14 days
  Arms: Intervention group
Dietary Supplement: Micro-encapsulated granules of sunflower oil (placebo) — Three times daily 4 grams of micro-encapsulated granules of sunflower oil, for a maximum of 14 days
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to investigate the possible effects of tributyrin supplementation in patients with a first episode of acute pancreatitis. The main question it aims to answer is:

• The effect of oral tributyrin supplementation on the plasma endotoxin level

Participants will be randomized between two groups: intervention and control group. They will receive:

- three times daily 4grams of micro-encapsulated granules of tributyrin, and the control group three times daily 4 grams of micro-encapsulated sunflower oil (i.e. placebo), for a total of 14 days

In total 92 adult patients with a first episode of acute pancreatitis will be included.

DETAILED DESCRIPTION:
Rationale: Acute pancreatitis (AP) is a common gastrointestinal disorder requiring acute hospitalization. Around 20% of patients that present with acute pancreatitis eventually develop severe complications such as (multiple) organ failure, (peri-) pancreatic necrosis, and secondary infections (i.e. infected necrosis, bacteraemia, pneumonia). The gut, especially the gut microbiome, is likely to play a role in development of infectious complications. Short-chain fatty acids (SCFAs) produced by the gut microbiota, such as butyrate, are known immunomodulators of the host response and exert local beneficial effects on the gut barrier and microbiota. Currently, there are no safe and effective therapies to mitigate disease severity that can be administered in the early phase of pancreatitis. We hypothesize that orally administered tributyrin, a pro-drug of butyrate, might beneficially influence disease progression in acute pancreatitis and may be useful as prophylaxis.

Objective: The main objective is to investigate the effect of oral tributyrin on plasma endotoxin in patients with acute pancreatitis after 3 days of treatment.

Study design: Phase IIa (Proof of concept) double-blind randomized placebo-controlled food supplement trial.

Study population: 92 adult patients with a first episode of acute pancreatitis.

Intervention: The intervention group receives three times daily 4g micro-encapsulated granules of tributyrin and the control group receives three times daily an equivalent volume of micro-encapsulated vegetable oil (i.e. placebo), for a total of maximum 14 days.

Main study parameters/endpoints: The primary endpoint is plasma endotoxin concentration after 3 days of tributyrin treatment. Secondary endpoints include toxicity, clinical outcomes, intestinal permeability, fecal SCFA concentrations, intestinal microbiota composition and systemic inflammatory response parameters (pulse, respiratory rate, temperature and white blood cell count).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The blood sampling at inclusion, and day 3 and 7 of treatment are preferably combined with regular blood sampling. Participants may experience minor discomfort from rectal swabs. Phase 1 studies with oral tributyrin conducted in patients with solid tumors did not report serious adverse events. However, there is a risk of unanticipated adverse events in our target population. An independent data safety and monitoring board (DSMB) will discuss all reported serious adverse events (SAE's).

ELIGIBILITY:
Inclusion Criteria:

* First episode of acute pancreatitis (AP)
* Able to read and/or understand the study procedures
* Able to give informed consent (or their legal representatives)
* <24 hours after diagnosis of AP
* <72 hours after onset of symptoms of AP

Exclusion Criteria:

* Pancreatitis due to endoscopic retrograde cholangiopancreatography (ERCP), malignancy or trauma
* Post-operative pancreatitis
* Intra-operative diagnosis
* Immunocompromised patients (history or current immunosuppressive treatment such as chemotherapy, radiotherapy, longer use of immunosuppressive medication or recent high doses, immunocompromised illness' such as AIDS, leukemia, lymphoma)
* Pregnancy and/or lactation
* Age <18 years old
* History of recurrent or chronic (MANNHEIM criteria25) pancreatitis (see Appendix 15.1 for definition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Plasma endotoxin levels | Measured 3 days after randomisation
  Plasma endotoxin levels

SECONDARY OUTCOMES:
Mortality | During the whole study period including follow-up of 90 days
  Occurence of death
Infectious complications | During the whole study period including follow-up of 90 days
  The occurence of infected pancreatic necrosis, bacteremia, pneumonia, urosepsis, and/or infected ascites
(New onset) transient/persistant (multiple) organ failure | During the whole study period including follow-up of 90 days
  The occurence of (new onset) transient/persistant (multiple) organ failure
Disease severity according to the revised Atlanta Classification | During the whole study period including follow-up of 90 days
  Disease severity according to the revised Atlanta Classification
(Peri-)pancreatic necrosis | During the whole study period including follow-up of 90 days
  The occurence of (peri)pancreatic necrosis
Length of hospital and/or ICU stay | During the whole study period including follow-up of 90 days
  Measured in days
The need (and number of) for surgical, endoscopic or radiologic interventions | During the whole study period including follow-up of 90 days
  The need (and number of) for surgical, endoscopic or radiologic interventions
Fecal and saliva microbiota and fecal metabolomics (i.e., SCFAs) analysis | During the whole study period including follow-up of 90 days
  Fecal and saliva microbiota and fecal metabolomics (i.e., SCFAs) analysis
Readmissions | During the whole study period including follow-up of 90 days
  The occurrence and number of readmissions
Systemic inflammatory response parameters (SIRS): pulse | During the initial admission
  Pulse measured in beats per minute
Systemic inflammatory response parameters (SIRS): respiratory rate | During the initial admission
  Respiratory rate measured in breaths per minute
Systemic inflammatory response parameters (SIRS): temperature | During the initial admission
  Temperature measured in degrees celsius
Systemic inflammatory response parameters (SIRS): white blood cell count | During the initial admission
  White blood cell count
Exocrine insufficiency | During the whole study period including follow-up of 90 days
  Exocrine insufficiency
Endocrine insufficiency | During the whole study period including follow-up of 90 days
  Endocrine insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: H. C. van Santvoort, dr. prof., Principal Investigator — St. Antonius Hospital
Locations (2):
- Netherlands (2):
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht

IPD SHARING:
Plan to Share IPD: No